CLINICAL TRIAL: NCT05937607
Title: The Effect of the Hand Massage Application on the Procedural Pain and State Anxiety of Women Undergoing Brachytherapy: A Parallel-Group Randomized Controlled Study
Brief Title: The Effect of the Hand Massage A Women Undergoing Brachytherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Dilek Efe Arslan, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 815/795
Record Dates: First submitted 2023-06-14; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Hand Massage
Keywords: Hand Massage; Pain; State Anxiety; Brachytherapy
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand massage (Experimental): hand massage was applied to the patients to receive intracavitary brachytherapy using lavender baby oil for three sessions of 10 minutes each, starting 5 minutes before the procedure.
  Interventions: Behavioral: Hand massage
- Control Group (No Intervention): The control group did not receive any intervention during the study period

INTERVENTIONS:
Behavioral: Hand massage — It is reported in the literature that the application should last 5-10 minutes on average to reduce acute pain, state anxiety, and provide physiological positive changes and relaxation in individuals during the procedure
  Arms: Hand massage

SUMMARY:
Background Gynecologic cancers are among the ten most common cancers among women. During brachytherapy, women can have pain and situational anxiety due to the treatment.

Methods This parallel-group randomized controlled study evaluated the effect of the hand massage practiced using baby oil, with lavender oil, on reducing operational pain and situational anxiety in women with brachytherapy. The study was completed with 36 patients. The treatment group included 18 patients, and the control group had 18. The data were collected through patient information form, visual analog scale, and state anxiety inventory. Before the brachytherapy, three sessions of hand massages, each lasting 10 minutes (5 minutes for each hand), were performed using baby oil with lavender. Data collection forms were repeated after each session. The control group received routine treatment. p<0.05 was accepted as significant.

DETAILED DESCRIPTION:
Therefore, the impact of hand massage applied with lavender baby oil on women with gynecologic cancer having brachytherapy for three sessions on the pain and state anxiety experienced during the intervention was evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* verbal communication
* to be at the age of 18 and above
* to be diagnosed with gynecologic cancer and receive BT three days a week regularly
* to be aware that she has a gynecologic cancer disease and to be a volunteer to participate in the study

Exclusion Criteria:

* the patients who had metastasis, bleeding or coagulation disorder
* received complementary and integrated treatment
* had edema or lesion on hand, had a psychiatric disease
* had communication problems
* did not want to have a massage
* were under general anesthesia during the intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | The scale was filled in the baseline
  VAS is a form including numbers and is used in rating pain. Patients mark their pain on a 10 cm ruler with painlessness 0 written on the left end and the most severe pain possible 10 on the right end. It is stated that VAS is more sensitive and dependable in pain severity measurement when compared to other one-dimensional scales

SECONDARY OUTCOMES:
State Anxiety Scale | The scale was filled in the baseline
  The state anxiety scale is sensitive to the evaluation of suddenly changing emotive reactions; it is a Likert-type scale including 20 questions. The reversed items in the scale were 1st, 2nd, 5th, 8th, 10th, 11th, 15th, 16th, 19th, and 20th items. High scores indicate elevated levels of anxiety, and low scores low levels of anxiety. The total score from the scale ranges between 20 and 80.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK EFE ARSLAN, PhD, Study Director — ERCİYES UNİVERSİTY
Locations (1):
- Dilek Efe Arslan, Kayseri, Talas, Turkey (Türkiye)